CLINICAL TRIAL: NCT01686841
Title: Pilot Clinical Trial Investigating the Effect of Cutaneous Cooling on Sebum Production
Brief Title: A Pilot Clinical Trial Investigating the Effect of Cutaneous Cooling on Sebum Production
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA12-003
Record Dates: First submitted 2012-09-12; First posted 2012-09-18 (Estimated); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Acne
Keywords: Cryolipolysis; Sebum
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- Sebum Reduction (Experimental): Subjects enrolled in the study were treated on the back with the Zeltiq System. Two sites on the upper back were selected as test sites and 1 site was used as a control.
  Interventions: Device: The Zeltiq System

INTERVENTIONS:
Device: The Zeltiq System — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis

SUMMARY:
To evaluate the safety and feasibility of reducing human sebum production using the ZELTIQ System.

DETAILED DESCRIPTION:
The study evaluated the use of the Zeltiq System to reduce sebum production on the upper back.

ELIGIBILITY:
Inclusion criteria

1. Male subjects >18 years of age and <25 years of age.
2. Subject has an average sebum output on their upper back of at least 20, as measured by the sebumeter
3. Subject has Fitzpatrick Skin Phototypes I-III (see Appendix A)
4. Willingness to participate in the study
5. Willingness to receive EXPERIMENTAL treatment
6. Informed consent agreement signed by the subject
7. Willingness to follow the treatment schedule and post treatment care requirements
8. Willingness to not use topical or systemic retinoids or antibiotics during the course of the treatment

Exclusion criteria

1. Subject has a history of isotretinoin use
2. Subject has an infection or other dermatologic condition (aside from acne) in the area to be treated
3. Subject has known cold sensitivity disorders including Raynaud's phenomena, cold urticaria, cryoglobulinemia, and cold induced hemoglobinuria
4. Presence of suntan in the area to be treated
5. Subject is immunosuppressed
6. Subject is unable to comply with treatment, home care or follow-up visits
7. Subject has a history of vitiligo
8. Subject has a history of keloid formation
9. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
10. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-08-16 (Actual); Primary Completion 2013-04-29 (Actual); Study Completion 2013-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rox Anderson, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 11 participants were enrolled and received treatment with the Zeltiq System using at -10C (Group 1) or -15C (Group 2). Each participant had 3 sites identified on their backs: 1 control site (no treatment) and 2 treatment sites.
Units Other Than Participants: Treatment Sites
Groups:
- Sebum ReductionTreatment Group 1 (-10C CoolSculpting Treatment): Participants were treated on 2 treatment sites on the upper back with the Zeltiq System using -10C and no treatment was received on 1 control site.
- Sebum Reduction Treatment Group 2 (-15C CoolSculpting Treatment): Participants were treated on 2 treatment sites on the upper back with the Zeltiq System using -15C and no treatment was received on 1 control site.
Period: Overall Study
Arm/Group | Sebum ReductionTreatment Group 1 (-10C CoolSculpting Treatment) | Sebum Reduction Treatment Group 2 (-15C CoolSculpting Treatment)
Started | 6; 18 Treatment Sites | 5; 15 Treatment Sites
Control Site | 6; 6 Treatment Sites | 5; 5 Treatment Sites
Treatment Sites | 6; 12 Treatment Sites | 5; 10 Treatment Sites
Completed | 6; 18 Treatment Sites | 5; 15 Treatment Sites
Not Completed | 0; 0 Treatment Sites | 0; 0 Treatment Sites

BASELINE CHARACTERISTICS:
Population: All enrolled participants treated with the Zeltiq System.
Groups:
- Sebum ReductionTreatment Group 1 (-10C CoolSculpting Treatment): Participants were treated on 2 treatment sites on the upper back with the Zeltiq System using -10C.
- Sebum Reduction Treatment Group 2 (-15C CoolSculpting Treatment): Participants were treated on 2 treatment sites on the upper back with the Zeltiq System using -15C.
- Total: Total of all reporting groups
Arm/Group | Sebum ReductionTreatment Group 1 (-10C CoolSculpting Treatment) | Sebum Reduction Treatment Group 2 (-15C CoolSculpting Treatment) | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 5 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Sebum Production in Treated Sites as Compared to Baseline Using Sebutape Measurements.
Description: Reduction of sebum production as measured by Sebutape at 2 weeks post-treatment. A 30% reduction of sebum production in a treated site compared to baseline Sebutape measurements will be considered clinically meaningful. Sebutape is an adhesive patch that acts as a passive collector of sebum. The gradual displacement of air in the pores of the microporous film changes its appearance. The size of the transparent area is a measure of the amount of sebum collected. All Sebutape measurements were performed in duplicate and the average of the two measurements was used for analysis. Results indicate the mean difference in Sebutape scores from baseline to 2 weeks post-treatment.
Time Frame: Baseline and 2 weeks post-treatment
Population: All enrolled participants presented here, as planned per protocol, by treatment received (-10C CoolSculpting Treatment or -15C CoolSculpting Treatment). Treatment Sites A and B were averaged.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Units Other Than Participants: treatment sites
Groups:
- Sebum Reduction Treatment Group 1A and 1B (-10C CoolSculpting Treatment): Participants were treated on 2 treatment sites on the upper back with the Zeltiq System using -10C; Participants were treated on site 1A of the upper back for a single 20 minute treatment with the Zeltiq System using -10C.
  Participants were treated on site 1B of the upper back for two 10 minute treatments with the Zeltiq System using -10C.
  Sites A and B were averaged.
- Sebum Reduction Treatment Group 1C (Control Site): Participants received no treatment to the control site 1C.
- Sebum Reduction Treatment Group 2A and 2B (-15C CoolSculpting Treatment): Participants were treated on 2 treatment sites on the upper back with the Zeltiq System using -15C; Participants were treated on site 2A of the upper back for a single 20 minute treatment with the Zeltiq System using -15C.
  Participants were treated on site 2B of the upper back for two 10 minute treatments with the Zeltiq System using -15C.
  Sites A and B were averaged.
- Sebum Reduction Treatment Group 2C (Control Site): Participants received no treatment to the control site 2C.
Arm/Group | Sebum Reduction Treatment Group 1A and 1B (-10C CoolSculpting Treatment) | Sebum Reduction Treatment Group 1C (Control Site) | Sebum Reduction Treatment Group 2A and 2B (-15C CoolSculpting Treatment) | Sebum Reduction Treatment Group 2C (Control Site)
Number analyzed (Participants) | 6 | 6 | 5 | 5
Number analyzed (treatment sites) | 12 | 6 | 10 | 5
Percent change from baseline | -10.9 (22.8) | 6.9 (11.1) | 7.8 (74.1) | 45.0 (103.7)

2. Primary Outcome: The Number of Unanticipated Adverse Device Effects (UADEs) Reported During the Study Period Will be Tabulated.
Description: The frequency of unanticipated adverse device effects (UADEs) reported throughout the study will be tabulated. Acceptance criteria: zero incidence of UADEs.
Time Frame: Time of enrollment through final 4-week follow-up visit
Population: All enrolled participants presented here, as planned per protocol, by treatment received (-10C CoolSculpting Treatment or -15C CoolSculpting Treatment).
Measure: Number; unit: events
Groups:
- Sebum Reduction Treatment Group 1 (-10C CoolSculpting Treatment): Participants were treated on 2 treatment sites on the upper back with the Zeltiq System using -10C.
Arm/Group | Sebum Reduction Treatment Group 1 (-10C CoolSculpting Treatment) | Sebum Reduction Treatment Group 2 (-15C CoolSculpting Treatment)
Number analyzed (Participants) | 6 | 5
events | 0 | 0

3. Secondary Outcome: The Number of Device- or Procedure-related Adverse Events Will be Tabulated.
Description: Device- or procedure related adverse events will be tabulated; side effects of treatment will be assessed.
Time Frame: Time of enrollment through the final 4-week follow-up visit
Population: All enrolled participants presented here, as planned per protocol, by treatment received (-10C CoolSculpting Treatment or-15C CoolSculpting Treatment).
Measure: Number; unit: events
Groups:
- Reduction Treatment Group 2 (-15C CoolSculpting Treatment): Participants were treated on 2 treatment sites on the upper back with the Zeltiq System using -15C.
Arm/Group | Sebum Reduction Treatment Group 1 (-10C CoolSculpting Treatment) | Reduction Treatment Group 2 (-15C CoolSculpting Treatment)
Number analyzed (Participants) | 6 | 5
events | 0 | 0

4. Secondary Outcome: Percent Change From Baseline of Sebum Production as Measured With Sebutape
Description: Sebum production will be measured using Sebutape at 72 hours, 1 week, and 4 weeks post-treatment. Sebutape is an adhesive patch that acts as a passive collector of sebum. The gradual displacement of air in the pores of the microporous film changes its appearance. The size of the transparent area is a measure of the amount of sebum collected. Sebutape measurements were performed in duplicate. The average of the two readings was used for analysis. Results are expressed in µg/cm² and correspond to the total amount of sebum collected on the film.
Time Frame: 72 hours post-treatment, 1 week post-treatment and 4 weeks post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from baseline
Units Other Than Participants: treatment sites
Arm/Group | Sebum Reduction Treatment Group 1A and 1B (-10C CoolSculpting Treatment) | Sebum Reduction Treatment Group 1C (Control Site) | Sebum Reduction Treatment Group 2A and 2B (-15C CoolSculpting Treatment) | Sebum Reduction Treatment Group 2C (Control Site)
Number analyzed (Participants) | 6 | 6 | 5 | 5
Number analyzed (treatment sites) | 12 | 6 | 10 | 5
percent change from baseline
  72 hours post treatment | 10.1 (27.3) | -9.7 (15.3) | 10.8 (26.3) | 26.7 (56.0)
  1 week post treatment | -17.0 (13.4) | -4.2 (10.2) | 46.0 (76.8) | 86.7 (110.2)
  4 weeks post treatment | 3.0 (26.2) | 6.9 (19.3) | 41.0 (58.9) | 43.3 (77.8)

5. Secondary Outcome: Number of Side Effect Events Post-treatment by Severity.
Description: All treatment sites (-10C vs -15C) were assessed for expected side effects of erythema, edema/swelling and dysesthesia at specific time points of the study. Treatment sites were scored on a 0 to 3 scale, with 0 = absent, 1 =minor, 2 = moderate and 3 = severe.
Time Frame: Post-treatment to 4-week final follow-up visit
Population: as for outcome 2
Measure: Number; unit: treatment sites
Units Other Than Participants: Treatment sites
Groups:
- Sebum Reduction Treatment Group 1A (-10C CoolSculpting Treatment): Participants were treated on 1 site of the upper back for a single 20 minute treatment with the Zeltiq System using -10C.
- Sebum Reduction Treatment Group 1B (-10C CoolSculpting Treatment): Participants were treated on 1 site of the upper back for two 10 minute treatments with the Zeltiq System using -10C.
- Sebum Reduction Treatment Group 1C (Control Site); Sebum Reduction Treatment Group 2C (Control Site): Participants received no treatment on the 1 control site.
- Sebum Reduction Treatment Group 2A (-15C CoolSculpting Treatment): Participants were treated on 1 site of the the upper back for a single 20 minute treatment with the Zeltiq System using -15C.
- Sebum Reduction Treatment Group 2B (-15C CoolSculpting Treatment): Participants were treated on 1 site of the upper back for two 10 minute treatments the Zeltiq System using -15C.
Arm/Group | Sebum Reduction Treatment Group 1A (-10C CoolSculpting Treatment) | Sebum Reduction Treatment Group 1B (-10C CoolSculpting Treatment) | Sebum Reduction Treatment Group 1C (Control Site) | Sebum Reduction Treatment Group 2A (-15C CoolSculpting Treatment) | Sebum Reduction Treatment Group 2B (-15C CoolSculpting Treatment) | Sebum Reduction Treatment Group 2C (Control Site)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 5
Number analyzed (Treatment sites) | 6 | 6 | 6 | 5 | 5 | 5
treatment sites
  Immediate post treatment erythema/purpura-absent | 0 | 0 | 6 | 0 | 0 | 5
  immediate post treatment erythema/purpura-minor | 1 | 1 | 0 | 0 | 0 | 0
  Immediate post treatment erythema/purpura -moderate | 5 | 5 | 0 | 5 | 5 | 0
  Immediate post treatment erythema/purpura - severe | 0 | 0 | 0 | 0 | 0 | 0
  Immediate post treatment edema/swelling-absent | 0 | 0 | 6 | 0 | 0 | 5
  Immediate post treatment edema-minor | 4 | 4 | 0 | 5 | 5 | 0
  Immediate post treatment treatment edema -moderate | 2 | 2 | 0 | 0 | 0 | 0
  immediate post-treatment edema- severe | 0 | 0 | 0 | 0 | 0 | 0
  Immediate post treatment dysesthesia =absent | 0 | 0 | 6 | 0 | 0 | 5
  Immediate post treatment dysesthesia -minor | 4 | 4 | 0 | 2 | 2 | 0
  Immediate post treatment dysesthesia -moderate | 2 | 2 | 0 | 3 | 3 | 0
  Immediate post treatment dysesthesia-severe | 0 | 0 | 0 | 0 | 0 | 0
  4 week F/U erythema/purpura-absent | 6 | 6 | 6 | 5 | 5 | 5
  4 week F/U erythema/purpura-minor | 0 | 0 | 0 | 0 | 0 | 0
  4 week F/U erythema/purpura- moderate | 0 | 0 | 0 | 0 | 0 | 0
  4 week F/U erythema/purpura -severe | 0 | 0 | 0 | 0 | 0 | 0
  4 week F/U edema- absent | 6 | 6 | 6 | 5 | 5 | 5
  4 week F/U edema -minor | 0 | 0 | 0 | 0 | 0 | 0
  4 week F/U edema-moderate | 0 | 0 | 0 | 0 | 0 | 0
  4 week F/U edema- severe | 0 | 0 | 0 | 0 | 0 | 0
  4 week F/U dysesthesia- absent | 6 | 6 | 6 | 5 | 5 | 5
  4 week F/U dysesthesia-minor | 0 | 0 | 0 | 0 | 0 | 0
  4 week F/U dysesthesia-moderate | 0 | 0 | 0 | 0 | 0 | 0
  4 week F/U dysesthesia-severe | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Any adverse event information was collected from the time of study enrollment through the 4-week post-treatment follow-up visit.
Description: The Safety Population consisted of all enrolled participants who received at least one study treatment. Data presented here, as planned per protocol, by treatment received (-10C CoolSculpting Treatment or -15C CoolSculpting Treatment).
Arm/Group | Sebum Reduction Treatment Group 1A (-10C CoolSculpting Treatment) | Sebum Reduction Treatment Group 1B (-10C CoolSculpting Treatment) | Sebum Reduction Treatment Group 1C (Control Site) | Sebum Reduction Treatment Group 2A (-15C CoolSculpting Treatment) | Sebum Reduction Treatment Group 2B (-15C CoolSculpting Treatment) | Sebum Reduction Treatment Group 2C (Control Site)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No